CLINICAL TRIAL: NCT00502619
Title: Pilot Study to Determine the Efficacy and Feasibility of a Structured Acupuncture and Treadmill Program to Treat Chronic Low Back Pain Patients to Improve Function, Exercise Capacity, and Pain Control.
Brief Title: Assessment of Acupuncture to Improve Function, Exercise Capacity, and Pain
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate recruitment of study subjects and inadequate retention.
Sponsor: VA Maryland Health Care System (U.S. Federal Agency)
Collaborators: Samueli Institute for Information Biology (Other)
Responsible Party: Robert Lavin, VA Maryland Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-27101; Samueli Institute: (Other Grant/Funding Number: 1 EA-0000060); Dept. of Defense IRB: (Other: A-13644.1)
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-07

CONDITIONS: Low Back Pain
Keywords: Low back pain; acupuncture; treadmill exercise
MeSH Terms: conditions — Low Back Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acupuncture plus Treadmill Exercise (Experimental): Acupuncture plus Treadmill Exercise
  Interventions: Procedure: Acupuncture; Other: Treadmill Exercise

INTERVENTIONS:
Procedure: Acupuncture — A specific regimen of acupuncture sites will be needled twice weekly for eight weeks and once weekly for a subsequent eight weeks.
Other: Treadmill Exercise — After the first four weeks of acupuncture treatments, subjects will initiate a three times per week treadmill program, which will continue for a total of 12 weeks in conjunction with the acupuncture treatments.

SUMMARY:
The purpose of this research proposal is to conduct a feasibility study to determine the viability a larger efficacy study of combined acupuncture treatments plus treadmill exercise to decrease pain, facilitate exercise, and improve function in Veterans with chronic low back pain (CLBP). To test this novel approach, subjects enrolled from a Veteran population at the Veteran Affairs Maryland Health Care System (VAMHCS) will undergo acupuncture plus low intensity treadmill walking exercise. Preliminary data regarding subject compliance, self-report of function, pain control, ambulatory activity, and exercise capacity will be collected to assess the response to this combined acupuncture/treadmill exercise protocol. Additionally, this study will determine the viability of this combined treatment paradigm for a larger study that will examine efficacy.

DETAILED DESCRIPTION:
Chronic non-malignant low back pain (CLBP) is very common. It is treated with diverse pharmacological and non-pharmacological therapies, including complementary and alternative pain treatments. Acupuncture has gained increasing acceptance among patients in the United States; however, the efficacy and duration of benefit of acupuncture treatments is often unknown, and prolonged utilization of these treatments is expensive. Successful acupuncture may provide an alternative to pain medications. Randomized studies have shown that exercise can produce long term benefits for individuals experiencing CLBP. Studies have also shown that acupuncture may be useful for the treatment of CLBP.

The purpose of the proposed research is to conduct a study to determine the feasibility of a larger efficacy study of acupuncture to decrease pain and facilitate exercise and function in Veterans with chronic low back pain (CLBP), in a Veteran population at the Veteran Affairs Maryland Health Care System (VAMHCS). To test this novel approach, subjects will undergo 16 weeks of treatment, consisting of acupuncture for 4 weeks followed by an overlapping period of 12 weeks of acupuncture plus low intensity treadmill walking exercise. Preliminary data will be collected to assess the improvement, if any, of: a) self-report of function, b) pain control, c) ambulatory activity, and d) exercise capacity. Additionally, this study will determine the viability of this combined treatment paradigm for a larger study that will examine efficacy.

Major objectives are to determine the rates of compliance for participation in this therapy of acupuncture plus low-intensity treadmill walking program, the completion rate of all treatment sessions and associated health assessment forms, as well as the challenges of recruitment. In addition, preliminary data to support the application for the larger pilot study will be obtained. The investigators' long-term research goal is to study this novel paradigm and its ability to reduce chronic low back pain.

The specific aims of the study are as follows:

Specific Objective 1. To determine whether individuals with CLBP receiving acupuncture plus treadmill exercise will exhibit superior improvement in function measured by Oswestry Disability Index II.

Specific Objective 2. To determine whether CLBP patients receiving acupuncture plus treadmill exercise will exhibit reduced pain scores measured by the Numeric Pain Intensity Rating Scale.

Specific Objective 3. To determine whether CLBP patients receiving acupuncture plus treadmill exercise will have improved home and community based ambulatory activity levels quantified by Step Activity Monitors (SAM).

Specific Objective 4. CLBP patients receiving acupuncture plus exercise will have greater gains in cardiovascular fitness levels measured by exercise testing with open circuit spirometry (V02 Max).

ELIGIBILITY:
Inclusion Criteria:

* Veterans eligible for this study are men or women between 25 and 65 years old with non-malignant low back pain greater than 6 months duration and pain scores greater than 4 (on a Numeric Pain Scale of 0 = No Pain and 10 = Worst Imaginable Pain) on most days out of the preceding month.
* Eligible subjects will also need to be able to tolerate 3 minutes walking at a rate of 0.5 miles per hour on a horizontal surface.

Exclusion Criteria:

* Inability to provide informed consent
* Diagnosis of dementia
* Severe depression (Beck Depression Inventory score > 30), suicidality, or untreated mental illness
* Severe anxiety (Beck Anxiety Inventory score > 30)
* Evidence of current substance abuse or alcoholism on the TICS
* Ongoing litigation related to the low back pain complaint
* Pregnancy or intent to become pregnant during time of study
* Ambulation requiring an assistive device
* Neurological, orthopedic, or other conditions impairing ambulation that would affect exercise safety
* Progressive neurological changes, altered sensation, or a history of cauda equina syndrome
* Pain below the knee that limits ambulation
* Lower extremity amputation proximal to the toes
* Low back pain problem requiring surgical intervention or impending surgery
* A history of lumbar vertebral fracture; and
* A history of prior lumbar surgery. Additional exclusion criteria include medical conditions that would affect an exercise program, such as rheumatologic, infectious, cardiac, peripheral vascular and pulmonary conditions, or ongoing cancer treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome measures are: (1) Numeric Pain Scale, (2) Oswestry Disability Index II, (3) fitness level determined by treadmill exercise, and (4) free-range ambulatory activity using step activity monitors. | 16 weeks

SECONDARY OUTCOMES:
Self-reports, including function, depression, anxiety, and sleep; a physical performance test battery. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Lavin, M.D., Principal Investigator — VA Maryland Health Care System
Locations (1):
- Baltimore VAMC, Baltimore, Maryland, United States